CLINICAL TRIAL: NCT06115473
Title: Intravenous Epinephrine Bolus for Prevention of Postintubation Collapse in Intensive Care Septic Patients Predicted by Shock Index.
Brief Title: Epinephrine to Prevent Postintubation Collapse in Shocked ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU R303/2023
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Shock
MeSH Terms: conditions — Shock | interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: : septic patients of either sex above 18 years of age, will need emergent intubation during ICU admission, shock index (SI) > 0.9.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E group for epinephrine (Active Comparator): In Group (E) patients will receive epinephrine prepared as 10 ml syringe filled with 10 ml of epinephrine 10 mcg/ml. prepared by drawing 1ml epinephrine 1mg ampule into 9 ml saline then discarding 9 ml and adding another 9 ml saline. now the investigators have 10 ml of epinephrine 10 mcg/ ml (1:100,000), then 10 µg will be given intravenously every 2-minute starting before intubation and continue during and after intubation for 4 times or until the systolic blood pressure (SBP) will be at least 90 mmHg or the mean arterial pressure (MAP) 65 mmHg or greater or after 4th dose of epinephrine and still hypotensive vasopressor (norepinephrine 30 ng /kg/min.) will be added or increased.
  Interventions: Drug: epinephrine
- Group (F) (Placebo Comparator): In Group (F) patients will receive IV bolus isotonic fluid 500 ml as it is yet the standard method used before intubation
  Interventions: Drug: isotonic fluid

INTERVENTIONS:
Drug: epinephrine — patients will receive epinephrine prepared as 10 ml syringe filled with 10 ml of epinephrine 10 mcg/ml. prepared by drawing 1ml epinephrine 1mg ampule into 9 ml saline then discarding 9 ml and adding another 9 ml saline. now the investigators have 10 ml of epinephrine 10 mcg/ ml (1:100,000), then 10 µg will be given intravenously every 2-minute starting before intubation and continue during and after intubation for 4 times or until the systolic blood pressure (SBP) will be at least 90 mmHg or the mean arterial pressure (MAP) 65 mmHg or greater or after 4th dose of epinephrine and still hypotensive vasopressor (norepinephrine 30 ng /kg/min.) will be added or increased.
  Arms: E group for epinephrine
Drug: isotonic fluid — patients will receive IV bolus isotonic fluid 500 ml
  Arms: Group (F)

SUMMARY:
Endotracheal intubation is a lifesaving procedure that is performed in various settings within the hospital or even in the pre-hospital field. However, it can result in serious hemodynamic complications, such as post-intubation hypotension (PIH) and cardiac arrest. Push-dose pressor (PDP) is common practice for rapid hemodynamic correction in post-intubation hypotension. In this study the investigators will use intravenous Epinephrine bolus for prevention of post intubation collapse in septic patients predicted by shock index in intensive care unit.

DETAILED DESCRIPTION:
* Type of Study: Randomized prospective comparative study.
* Study Setting: Ain Shams University Hospitals at Intensive care units department. • Study Period: 4 months.
* Study Population: -Inclusion Criteria: septic patients of either sex above 18 years of age, will need emergent intubation during ICU admission, shock index (SI) > 0.9.

Exclusion Criteria: patient's family refusal, age <18, pregnant, Patients with tachyarrhythmias, traumatic patients, patient with shock index <0.9, ischemic heart patients, any comorbidities contraindicated to take epinephrine and allergic to epinephrine will be excluded from the study. • Sampling Method: Study will include (44) patients who fulfill all the points in the inclusion criteria will be randomized into 2 equal groups, each consisting of (22) patients, namely group (E) and group (F). • Sample Size: 44 patients.

• Ethical Considerations: Approval of the Ethical Committee and written informed consent from all participants' legal guardians will be obtained after explanation. • Study Procedures: Push-dose epinephrine will be prepared (following mixing instructions) and administered via large bore (14-18 gauge) peripheral intravenous (IV) access.

(44) Patients will randomly be assigned into two groups, (E group for epinephrine n= 22, F group for IV bolus isotonic fluid n=22). Randomization will be done using sequentially numbered, opaque, sealed envelopes containing computer generated random allocations.

In Group (E) patients will receive epinephrine prepared as 10 ml syringe filled with 10 ml of epinephrine 10 mcg/ml. prepared by drawing 1ml epinephrine 1mg ampule into 9 ml saline then discarding 9 ml and adding another 9 ml saline. now the investigators have 10 ml of epinephrine 10 mcg/ ml (1:100,000), then 10 µg will be given intravenously every 2-minute starting before intubation and continue during and after intubation for 4 times or until the systolic blood pressure (SBP) will be at least 90 mmHg or the mean arterial pressure (MAP) 65 mmHg or greater or after 4th dose of epinephrine and still hypotensive vasopressor (norepinephrine 30 ng /kg/min.) will be added or increased. In Group (F) patients will receive IV bolus isotonic fluid 500 ml as it is yet the standard method used before intubation.

Blood pressure, heart rate, oxygen saturation will be measured before intubation and every 5 minutes for 30-minute, lactate will be measured at intubation and 6-hour postintubation. Incidence of arrythmia will be recorded.

Primary intention will be incidence of cardiac arrest during intubation or sever hypotension (decrease > 20% of baseline mean arterial blood pressure) (Bijker et al, 2007).

Secondary intention will be incidence of arrythmias, bradycardia (heart rate < 50/minute), increased lactate, need for or increase dose of postintubation vasopressor (norepinephrine 30 ng /kg/min.) and decreased oxygen saturation.

Sample size: Data collected will be analyzed using PASS 15 program for sample size calculation, setting power 80% and alpha error at 0.05 and according to "panchal et al, 2015 ", the expected increase in SBP and DBP in epinephrine group is about 25%. Assuming no change in control group, sample size 22 patients per group will be needed to detect the difference between groups.

Statistical analysis: will be performed using computer software statistical package for the social science (SPSS, version 20; SPSS Inc., Chicago, Illinois, USA). Description of Quantitative (numerical) variables will be performed in the form of mean ± SD. Description of the qualitative (categorical) data will be performed in the form of numbers of cases and percent. Error bars represent 95% confidence interval. ANOVA test and chi-square tests will be used for comparison among different times in the same group in quantitative data. Significance level will be set at P-value of 0.05 or less, and P-value of 0.01 or less will be considered highly significant.

ELIGIBILITY:
Inclusion Criteria:

* septic patients of either sex above 18 years of age, will need emergent intubation during ICU admission, shock index (SI) > 0.9.

Exclusion Criteria:

* patient's family refusal, age <18, pregnant, Patients with tachyarrhythmias, traumatic patients, patient with shock index <0.9, ischemic heart patients, any comorbidities contraindicated to take epinephrine and allergic to epinephrine will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
incidence of cardiac arrest during intubation | during and till 30 minutes after intubation
  cardiac arrest
sever hypotension | during and till 30 minutes after intubation
  decrease > 20% of baseline mean arterial blood pressure

SECONDARY OUTCOMES:
incidence of arrythmias | during and till 30 minutes after intubation
  arrythmias
bradycardia | during and till 30 minutes after intubation
  heart rate < 50/minute
increased lactate | lactate will be measured 1 hour after intubation
  more than base line
need for or increase dose of postintubation vasopressor | during and till 30 minutes after intubation
  norepinephrine 30 ng /kg/min.
decreased oxygen saturation | during and till 30 minutes after intubation
  less than 90%

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals at Intensive care units department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided